CLINICAL TRIAL: NCT05586087
Title: Effects of an High-Speed Resistance Training Program on Health Parameters in Independent Older Adults: a Longitudinal Study
Brief Title: High-Speed Resistance Training Program in Independent Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: Polytechnic Institute of Rio Maior (Other); Comprehensive Health Research Center (Other); Foundation for Science and Technology, Portugal (Other); Life Quality Research Center - CIEQV (Unknown)
Responsible Party: Principal Investigator, Alexandre Duarte Martins, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Idade Activa
Record Dates: First submitted 2022-10-04; First posted 2022-10-19 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Old Age; Atrophy; Aging
Keywords: Aging; Older adults; Resistance training; Velocity-based training; Health outcomes; Phase Angle; Gait Variability
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants perform a 16-week of High-Speed Resistance Training program.
  Interventions: Other: Experimental group
- Control group (No Intervention): Participantes continued their usual activity without engaging in any strength training or beginning a new exercise program during the study.

INTERVENTIONS:
Other: Experimental group — The High-Speed Resistance Training program has 16 weeks, with three sessions per week with 50-60min, each session being comprised of five-six exercises, two-three sets, and six-ten reps/exercise. The intensity is gradually increased after each session in accordance with the movement velocity (>1.3 to 0.75 m/s) representing approximately 20% to 60% of one repetition maximum. Participants execute the exercises rapidly and explosively making all repetitions for each shortening phase (concentric phase) performed as quickly as possible with the lengthening phase of the muscle (eccentric phase) being controlled for 2-3 s. The velocity of the concentric phase in each exercise is monitored through a BEAST™ sensor (Beast Technologies, Brescia, Italy).
  Arms: Experimental group

SUMMARY:
The aims of the present investigation are: a) to determine the effects of a 16-weeks high-speed resistance training program on health parameters in independent older adults; and b) to verify the durability of the effects after 6 and 12 months after the intervention.

DETAILED DESCRIPTION:
The present investigation will last a total of 18 months. More specifically, Two weeks for initial assessments, then the 16-weeks training program. After that, there will be a 1-year follow-up.

Regarding the training program, it consists in a high-speed resistance training program of 16-weeks, with three sessions per week (Mondays, Wednesdays, and Fridays) of 50-60min, each session being comprised of five-six exercises, two-three sets, and six-ten reps/exercise. The following exercises are used during the intervention period in pneumatic machines: incline bench press, squat in multipower or with dumbbell, leg extension, seated low row, leg press, calf raise, chest fly and lat pull down.

The intensity is gradually increased after each session in accordance with the movement velocity (>1.3 to 0.75 m/s) representing approximately 20% to 60% of one repetition maximum. Participants execute the exercises rapidly and explosively making all repetitions for each shortening phase (concentric phase) performed as quickly as possible with the lengthening phase of the muscle (eccentric phase) being controlled for 2-3 s. The velocity of the concentric phase in each exercise is monitored through a BEAST™ sensor (Beast Technologies, Brescia, Italy).

Participants unavailable to participate in the intervention period will be allocated to the control group. These participants continue their usual activity without engaging in any resistance training or beginning a new exercise program during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders;
* Aged 65 years old or more;
* Can walk and perform daily tasks independently and autonomously.

Exclusion Criteria:

* People with cognitive impairment;
* People with neurodegenerative diseases;
* People with diabetes disease;
* People with heart/respiratory pathology or use of pacemakers;
* People with musculoskeletal injuries in the 6 months before the study;
* People with active oncology disease;
* People with an uncontrolled hypertension (>90 mmHG; >150 mmHg);
* People participate in other supervised exercise program;
* Paeople who refuse to sign the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Phase angle from bioelectrical impedance | 18 months
  Changes related to cellular health assessed by In Body S10 after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Gait Variability | 18 months
  Changes related to gait variability by Phypox after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.

SECONDARY OUTCOMES:
Body Composition - Muscle mass; Fat Mass; Body Water. | 18 months
  Changes related to muscle mass, fat mass and body water assessed by In Body S10 and DXA after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Bone Densitometry - Whole-body BMC and BMD and dominant femoral neck BMC and BMD. | 18 months
  Changes related to bone quality assessed by DXA after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Heart Rate Variability | 18 months
  Changes related to autonomous nervous system assessed by Kubios HRV after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Physical Function | 18 months
  Changes related to physical function assessed by four functional fitness tests, namely 30s chair-stand; timed-up & go test; ball throw and 6 min walk test after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Muscle strength | 18 months
  Changes related to Muscle strength assessed by handgrip test (both sides) and isokinetic dynamometer evaluation (both sides) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Postural control | 18 months
  Changes related to postural control assessed in two conditions (with one foot on the ground and both feet on the ground) by an force platform Add-on (Plux) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Falls Efficacy Scale - International (FES-I) | 18 months
  Changes related to the level of concern about falling during social and physical activities inside and outside the home through a scale (FES-I) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
International Physical Activity Questionnaire (IPAQ) | 18 months
  Changes related to the levels of physical activity through a scale (IPAQ) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
Mini-Mental State Examination | 18 months
  Changes related to the cognitive impairment (problems with thinking, communication, understanding and memory) through a scale (MMSE) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.
The 36-Item Short Form Survey (SF-36) | 18 months
  Changes related to the health status through a scale (SF-36) after a 16-weeks high-speed resistance training program and after 6 and 12 moths of the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Health, School of Health and Human Development, University of Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duarte Martins A, Paulo Brito J, Fernandes O, Oliveira R, Goncalves B, Batalha N. Effects of a 16-week High-Speed Resistance Training program on body composition in community-dwelling independent older adults: A clinical trial. Clin Nutr ESPEN. 2024 Oct;63:84-91. doi: 10.1016/j.clnesp.2024.06.010. Epub 2024 Jun 20. PMID 38935496